CLINICAL TRIAL: NCT01052766
Title: The Use of Breathing Synchronized PET/CT Scans for the Detection of Malignant Lung and Liver Lesions and Assessment of Tumor Glycolysis
Brief Title: Breathing Synchronized PET/CT Scans for the Detection of Malignant Lung & Liver Lesions and Assessment of Tumor Glycolysis
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-134
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Last update posted 2012-03-16 (Estimated); Status verified 2012-03

CONDITIONS: Lung Cancer; Non-small Cell Lung Cancer
Keywords: lung cancer; PET Scan; CT Scan; BH-PET scan; 09-134
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

ARMS (1):
- PET/CT and BH PET/CT (Experimental): In collaboration with the Department of Radiation Oncology and the Interventional Radiology Service, patients with lung or liver cancer or lung or liver metastases in whom FDG PET/CT is part of the clinical standard of care for disease evaluation and response assessment will be enrolled in this study. We will perform a clinical PET/CT and BH PET/CT (for two bed positions covering the entire chest) prior to, and again 1-2 weeks after SBRT or RFA. This early time point is chosen because a few weeks after the completion of treatment, acute radiation injury in the lung begins and will likely be detectable as abnormal uptake on follow-up PET imaging making it difficult to assess tumor recurrence.
  Interventions: Procedure: PET/CT and BH PET/CT

INTERVENTIONS:
Procedure: PET/CT and BH PET/CT — First, fiducial markers will be placed and taped on the patient's lower chest/upper abdomen. This will allow for monitoring of chest motion during breathing. A BH-CT scan will then be acquired with clinical CT scan parameters used in nuclear medicine. A BH-PET scan (acquisition time: 6 min per bed position) will follow the BH-CT scan. BH-PET images will cover the whole thorax, which, on average, corresponds to 1-3 PET FOV's (~15 cm/FOV). Data for these 1-3 bed positions are acquired to cover the entire thorax. There will be no additional radiotracer injection for the BH-PET scan.

SUMMARY:
In this particular study the physicians want to use a new technique of how they obtain the PET/CT pictures. It is called breath-hold (BH) PET/CT". As the name suggests, they will ask the patient to hold their breath for about 20-30 seconds, and only during that time will they obtain pictures. This is repeated several times. In contrast to the standard PET/CT scan, they expect less "blurring" of the pictures, so that they can see the tumor better and measure the uptake of radioactive sugar in the tumor better and more reliably. Basically, this is the difference between taking pictures of a runner as compared to taking pictures of a person standing still. Since PET images need to be obtained over several minutes and people can not hold their breath for this extended time, we break the procedure into several cycles of 20-30 seconds (or longer, if possible) and then add all the "frozen" pictures in the end into one. They want to know if BH PET/CT scan measure changes in the cancer during therapy (i.e., from the baseline scan before therapy to the follow up scan at within 4 weeks later).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients with early stage biopsy-proven lung cancer or patients with lung or liver metastases from any primary cancer (metastatic disease proven by biopsy, or clearly established clinically and by imaging studies who are being treated with stereotactic body radiotherapy (SBRT)or an ablation will be eligible.
* Patient has at least one lesion ≥ 1cm in size.
* Signed informed consent

Exclusion Criteria:

* Pregnant women are ineligible.
* Patients who are unable to follow breathing instructions either due to language difficulties or hearing impairment This will be determined either by one of the consenting individuals when they approach the patient to ask for informed consent or prior to acquisition of the clinical PET/CT.
* Patients who are too ill to hold their breath.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2010-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
To investigate whether BH-PET scan improves detectability of the lung & liver lesions seen on breath-hold CT scans as compared to their detectability on standard clinical PET scan. | 2 years

SECONDARY OUTCOMES:
To compare the magnitude of changes in SUV between pre and post therapy pet scans done as either standard clinical PET/CT or BH PET/CT. | 2 years
To investigate whether the correlation between change in SUV and the lesion response on follow-up scan (3 months) is different for standard clinical PET/CT versus BH scan. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Heiko Schoder, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm